CLINICAL TRIAL: NCT02809716
Title: High Definition Single Cell Analysis in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 3C-15-4; NCI-2016-00736 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-15-4 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-06-19; First posted 2016-06-22 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Carcinoma in the Liver; Stage IV Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (blood and tumor tissue collection): Patients undergo collection of blood collection 1 week prior surgery, before and after surgery on the same day, and 1 week and 3 months after surgery. Patients also undergo and tissue collection during the surgery. Blood and tissue samples are processed for high definition single cell analysis including, whole-genome CNV profiles, protein expression, and cell morphology.
  Interventions: Other: Biomarker Analysis; Other: Cytology Specimen Collection Procedure

INTERVENTIONS:
Other: Biomarker Analysis — Correlative studies
Other: Cytology Specimen Collection Procedure — Undergo collection of blood and tissue samples
  Other Names: Cytologic Sampling

SUMMARY:
This research clinical trial studies high definition single cell analysis in blood and tissue samples from patients with colorectal cancer which has spread to the liver. High definition single cell analysis allows doctors to study the properties of cancer cells that are sometimes found in the blood of patients and to determine how the genes and proteins in them may change over time. Studying samples from patients with colorectal cancer in the laboratory may help doctors learn more about how cancer spreads, as well as how to predict the disease outcomes in patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the level of correlation between solid tumor touch preparations and liquid biopsies (circulating tumor cells [CTCs]) from patients with surgically resected colorectal cancer (CRC) metastases to the liver using single-cell high-content analysis, including gene copy number variation (CNV) and to establish one or more bio-signatures that represent the liquid and solid biopsy correlation for each patient and for the patient population.

SECONDARY OBJECTIVES:

I. To demonstrate the technical validity and reproducibility of the bio-signatures by comparing the two pre-resection liquid biopsy samples drawn one week prior to and on the day of surgery.

TERTIARY OBJECTIVES:

I. Compare biosignatures between pre-surgical and post-surgical blood samples. II. Compare biosignatures between resected metastatic liver tumor tissue, primary colon tumor tissue (if available), and pre-surgical blood samples.

III. Compare biosignatures between blood samples prior to resection with those obtained after resection and at the time of recurrence.

OUTLINE:

Patients undergo blood collection 1 week prior surgery, before and after surgery on the same day, and 1 week and 3 months after surgery. Patients also undergo tissue collection during the surgery. Blood and tissue samples are processed for high definition single cell analysis including whole-genome CNV profiles, protein expression, and cell morphology.

After completion of study, patients are followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Metastatic colorectal adenocarcinoma to the liver (hepatic mCRC)

  * Synchronous or metachronous
  * Solitary or multifocal
  * Concurrent abdominal lymph node metastasis is allowable
* Hepatic mCRC deemed surgically resectable by the study team with plans to undergo surgery
* Has not received any systemic chemotherapy for at least 21 days prior to scheduled hepatic resection

Exclusion Criteria:

* Non-adenocarcinoma metastatic colorectal cancer (e.g. neuroendocrine carcinoma); mucinous component is permitted
* Metastatic CRC that involves organ(s)/tissue(s) other than abdominal lymph nodes and/or liver
* Has received any systemic chemotherapy within 21 days prior to scheduled hepatic resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic CRC with single- and multi-focal hepatic lesions scheduled for resection (metastatectomy)
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
HD-SCA liquid biopsy biosignatures assessed by cell morphology, protein expression, and whole genome CNV profiles | Up to 2 years
  Biosignatures will be compared between cells from tumor tissue within the same patient, cells from blood samples within the same patient, cells from tumor tissue and blood samples within the same patient, cells from tumor tissue and blood samples across different patients. Upon these comparisons, biosignatures will be established which represent liquid and solid biopsy correlations for each patient and for the patient population. Descriptive statistics will be used to determine means, correlations, and variability of biosignatures between different specimens and time points, and within and acr
HD-SCA solid tumor biosignatures assessed by cell morphology, protein expression, and whole genome CNV profiles | Up to 2 years
  Biosignatures will be compared between cells from tumor tissue within the same patient, cells from blood samples within the same patient, cells from tumor tissue and blood samples within the same patient, cells from tumor tissue and blood samples across different patients. Upon these comparisons, biosignatures will be established which represent liquid and solid biopsy correlations for each patient and for the patient population. Descriptive statistics will be used to determine means, correlations, and variability of biosignatures between different specimens and time points, and within and acr

SECONDARY OUTCOMES:
HD-SCA biosignatures in pre-resection liquid biopsy samples assessed by cell morphology, protein expression, and whole genome CNV profiles | Up to day 1 of surgery
  The technical validity and reproducibility of the biosignatures will be demonstrated by comparing two pre-resection liquid biopsy samples. This reflects a change in the timing of specimen collection from the original protocol. Descriptive statistics will be used to determine means, correlations, and variability of biosignatures between different specimens and time points, and within and across patients.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kuhn, Principal Investigator — University of Southern California
Locations (6):
- United States (6):
  - Scripps Cancer Center, La Jolla, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas